CLINICAL TRIAL: NCT05110521
Title: Impact of a Nurse Mentorship and Digital Health Package Intervention for Maternal and Newborn Health in Kenya: A Cluster Randomized Controlled Trial
Brief Title: Evaluation of a Nurse Mentorship and Digital Health Package Intervention in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Innovations for Poverty Action (Other); Jacaranda Health (Other)
Responsible Party: Principal Investigator, Jessica Cohen, Associate Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB21-1013
Record Dates: First submitted 2021-10-25; First posted 2021-11-08 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Quality of Care
Keywords: maternal and newborn health; quality of care; mentorship; mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (PROMPTS and MENTORS offered) (Experimental): Health facilities randomized into the Intervention Arm will be offered the MENTORS program, which trains in-facility nurse-mentors to provide health workers with training and mentorship on aspects of basic and emergency obstetric and newborn care. At health facilities in the intervention arm, patients attending antenatal care clinics will be offered the PROMPTS program, which is a digital health platform that connects mothers with information, advice and referrals to care.
  Interventions: Behavioral: PROMPTS; Behavioral: MENTORS
- Control (Routine Care/No PROMPTS or MENTORS OFFERED) (No Intervention): In the control arm, neither the PROMPTS program nor the MENTORS program will be offered during the study period.

INTERVENTIONS:
Behavioral: PROMPTS — PROMPTS is a two-way Short Message Service (SMS) digital health platform that connects mothers with information, advice and referrals to care during the prenatal and postnatal period. The platform also collects information from women on care experience that is reported back to maternity facilities.
  Arms: Intervention (PROMPTS and MENTORS offered)
Behavioral: MENTORS — MENTORS is a program in which in facility nurse-mentors are trained and supported to offer training to nurses, midwives and other maternity facility staff on aspects of basic and emergency obstetric and newborn care.
  Arms: Intervention (PROMPTS and MENTORS offered)

SUMMARY:
The investigators will conduct a cluster randomized controlled trial in maternity facilities in Kenya to evaluate the impact of a maternal and neonatal health package intervention on patient and provider outcomes. This package intervention includes two programs: PROMPTS, a digital health platform for mothers aimed to improve knowledge and health behaviors and increase care-seeking behavior at the right time and place, and MENTORS, a facility-based program aimed to increase and sustain providers' knowledge and skills in basic and emergency obstetric and newborn care. Facilities will be randomized into a treatment group that receives the package or a control group that receives usual care. Patient outcomes include health knowledge, health behaviors and health care utilization in the prenatal and postnatal period; provider outcomes include knowledge and quality of care.

DETAILED DESCRIPTION:
This study is designed as a parallel arm cluster randomized controlled trial (RCT). Randomization of the intervention package will occur at the facility level. The investigators will randomize 40 facilities across 8 counties into either the intervention or control group.

Data will be collected at multiple points during the study period. Facility baseline data collection will occur over a one month period in each facility. Baseline data collection will include a facility assessment, maternity register data extraction and health worker interviews.

In order to evaluate the PROMPTS component of the intervention, the investigators will enroll a cohort of women during baseline facility data collection that will be followed through their pregnancy, delivery and postpartum period. The investigators will recruit pregnant women attending study clinics for antenatal care during the baseline data collection period. They will be surveyed by phone twice in the follow-up period: once in the last month of pregnancy and again at 7- to 8-weeks postpartum. Women enrolled from the intervention facilities will be offered the PROMPTS intervention immediately after the baseline survey.

The facility-based endline data collection will occur 4-5 months after the end of baseline and will last for 1-2 months in each facility. The facility-based endline data collection will include register data extraction, health worker interviews, and observations of quality of care during labor and delivery.

A process evaluation will be conducted using administrative program data collected by Jacaranda Health to monitor intervention implementation within the treatment facilities.

After the endline, facilities in the control group will also be offered the intervention.

ELIGIBILITY:
Inclusion Criteria for Health Facilities:

* have at least 50 normal vaginal deliveries per month on average
* have at most 400 normal vaginal deliveries per month on average
* are owned by the government or a faith-based organization
* have no potentially confounding ongoing research or quality-improvement programs at the time of selection (especially mentorship or mHealth programs).

Inclusion Criteria for Participants of Provider Surveys:

* nurses or midwives
* provide delivery care in the study facility
* have no plan to move to a different facility in the next 6 months (baseline only).

Inclusion Criteria for Participants of PROMPTS Surveys:

* at least 15 years old
* have access to a mobile phone
* are at least 16 weeks pregnant or in Month 5, 6, 7, 8, and 9 of pregnancy.

Inclusion Criteria for Participants of Delivery Observations:

* at least 15 years old
* are admitted for labor and delivery at the maternity ward

Exclusion Criteria for Participants of Delivery Observations:

* are presenting for conditions other than labor and delivery (e.g., patients admitted for prenatal observation or complications from abortion)
* are immediately transferred to another hospital.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10992 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Quality of routine maternity care, measured by delivery observation | assessed from patient admission to up to 1 hour post the delivery of the placenta approximately 6 months after intervention initiation
  A ratio based on a 20-item index that measures essential actions providers must perform during the course of labor and delivery (Tripathi et al., 2015). The total score is calculated as the fraction of 20 items weighted equally, yielding a range of 0 to 1, with higher scores indicating better quality of maternal care.
Provider knowledge on obstetric and newborn care, measured by provider survey | assessed approximately 6 months after intervention initiation
  A continuous variable based on the answers to 10 questions on normal labor, infection prevention and control, preeclampsia and eclampsia, newborn care, postpartum hemorrhage, and shoulder dystocia.
Patient knowledge on danger signs, measured by patient survey | assessed in the last month of pregnancy (prenatal danger signs) and between 7 - 8 weeks postpartum (neonatal and postpartum danger signs)
  A ratio based on questions that ask whether a respondent would seek medical care immediately in response to serious prenatal, neonatal, and postpartum danger signs. Each question is scored according to whether a participant chooses the correct response (i.e., whether to visit a hospital/call a doctor or not in response to a serious health condition). The total score is calculated as the share of the times the respondent correctly identifies the need to seek medical care immediately.
Care seeking in response to severe danger signs, measured by patient survey | assessed in the last month of pregnancy (prenatal danger signs) and between 7 - 8 weeks postpartum (neonatal and postpartum danger signs)
  A binary variable based on a series of questions that measure whether a respondent sought any medical advice or treatment for a healthcare provider in response to severe prenatal, postnatal, and neonatal danger signs. The variable is coded to one if respondent sought advice or treatment for at least one danger sign.
Postnatal care for mom within six weeks postpartum, measured by patient survey | assessed at 7 - 8 weeks postpartum
  a binary variable equal to 1 if there was at least 1 postnatal visit within six weeks postpartum AND mom's own health was discussed during the postnatal care visit
Number of antenatal care visits, measured by patient survey | assessed between 7 - 8 weeks postpartum
  a continuous variable for the total number of antenatal care visits during the entire pregnancy
Quality of care for management of neonatal resuscitation, measured by simulation exercise | assessed approximately 6 months after intervention initiation
  A continuous variable based on providers' actions in a simulation exercise for neonatal resuscitation. Each question is scored according to whether a provider performs the correct step for neonatal resuscitation. The total score is calculated as the sum of all questions. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Quality of care for management of maternal and neonatal complications, measured by delivery observation | assessed from patient admission to up to 1 hour post the delivery of the placenta approximately 6 months after intervention initiation
  A continuous variable based on essential actions providers should perform to manage maternal and neonatal complications, including postpartum hemorrhage, pre-eclampsia/eclampsia, neonatal resuscitation, and shoulder dystocia. Score is calculated as the fraction of total items applicable to each case. The total score has a range of 0 to 1, with higher scores indicating better quality of care.
Quality of care for infection prevention, measured by delivery observation | assessed from patient admission to up to 1 hour post the delivery of the placenta approximately 6 months after intervention initiation
  A continuous variable based on a series of questions that measure whether infection prevention and control procedures are performed during labor and delivery. Individual item is assigned a score equal to 1 if an action is done.
Quality of care for partograph completion, measured by delivery observation | assessed from patient admission to up to 1 hour post the delivery of the placenta approximately 6 months after intervention initiation
  A continuous variable based on a series of questions that measure whether progress of labor is plotted appropriately on the partograph. Individual item is assigned a score equal to 1 if an action is done.
Provider motivation and satisfaction, measured by provider survey | assessed approximately 6 months after intervention initiation
  A continuous variable based on 11 questions that measure health workers' motivation adapted from a scale validated in Kenya (Mbindyo et al, 2009). Individual questions are scored using a 1-to-5 LIkert scale. The total score is calculated as the sum of all items (with a few items reverse coded).
Patient treatment during labor and delivery, measured by delivery observation | assessed from patient admission to up to 1 hour post the delivery of the placenta approximately 6 months after intervention initiation
  A continuous variable based on a series of questions that measure aspects of mistreatment during labor and delivery: interpersonal abuse scale, exams & procedures index, and unsupportive birth environment (Berger et al., 2021). Individual items are scored to 1 if observed.
Respectful maternity care during last antenatal care visit, measured by patient survey | assessed between 36 - 42 weeks' gestation
  A binary variable equal to one if a patient felt she was treated with respect during her last antenatal care visit.
Disrespect in care during delivery, measured by patient survey | assessed between 7 - 8 weeks postpartum
  An ordinal variable based on to what extent a patient was abused or treated in a way that made her feel humiliated/disrespected during her delivery.
Severe morbidity and mortality, measured by delivery observation and document review | assessed at approximately 6 months after intervention initiation
  A composite binary variable that measures whether a woman or her baby had any severe maternal complication (including severe postpartum hemorrhage, severe pre-eclampsia, eclampsia, severe systemic infection or sepsis, and uterine rupture), neonatal complication (including asphyxia), maternal mortality, and perinatal mortality (including stillbirth and newborn death). The value of this outcome will be 1 if a woman or her baby had at least one complication listed or died.
Medical advice/treatment seeking during pregnancy, measured by patient survey | assessed between 36 - 42 weeks' gestation
  A binary variable that measures whether a participant sought advice or treatment from a healthcare professional in the past month
Medical advice/treatment seeking for baby's health postpartum, measured by patient survey | assessed between 7 - 8 weeks postpartum
  A binary variable that measures whether a participant sought advice or treatment from a healthcare professional since she left the hospital after delivery for her baby's health
Medical advice/treatment seeking for mom's health postpartum, measured by patient survey | assessed between 7 - 8 weeks postpartum
  A binary variable that measures whether a participant sought advice or treatment from a healthcare professional since she left the hospital after delivery for her own health
Care seeking in response to severe antenatal danger signs, measured by patient survey | assessed between 36 - 42 weeks' gestation
  A binary variable based on a series of questions that measure whether a respondent sought any medical advice or treatment for a healthcare provider in response to severe prenatal danger signs.The variable is coded to one if respondent sought advice or treatment for at least one danger sign.
Care seeking in response to severe postnatal danger signs, measured by patient survey | assessed between 7 - 8 weeks postpartum
  A binary variable based on a series of questions that measure whether a respondent sought any medical advice or treatment for a healthcare provider in response to severe postnatal danger signs. The variable is coded to one if respondent sought advice or treatment for at least one danger sign.
Care seeking in response to severe neonatal danger signs, measured by patient survey | assessed between 7 - 8 weeks postpartum
  A binary variable based on a series of questions that measure whether a respondent sought any medical advice or treatment for a healthcare provider in response to severe neonatal danger signs. The variable is coded to one if respondent sought advice or treatment for at least one danger sign.
Patient knowledge on prenatal danger signs, measured by patient survey | assessed between 36 - 42 weeks' gestation
  A ratio based on questions that ask whether a respondent would seek medical care immediately in response to serious prenatal danger signs. Each question is scored according to whether a participant chooses the correct response (i.e., whether to visit a hospital or not in response to a health condition). The total score is calculated as the share of the times the respondent correctly identifies the need to seek medical care immediately..
Patient knowledge on postnatal danger signs, measured by patient survey | assessed between 7 - 8 weeks postpartum
  A ratio based on questions that ask whether a respondent would seek medical care immediately in response to serious postpartum danger signs. Each question is scored according to whether a participant chooses the correct response (i.e., whether to visit a hospital or not in response to a health condition). The total score is calculated as the share of the times the respondent correctly identifies the need to seek medical care immediately.
Patient knowledge on neonatal danger signs, measured by patient survey | assessed between 7 - 8 weeks postpartum
  A ratio based on questions that ask whether a respondent would seek medical care immediately in response to serious neonatal danger signs. Each question is scored according to whether a participant chooses the correct response (i.e., whether to visit a hospital or not in response to a health condition). The total score is calculated as the share of the times the respondent correctly identifies the need to seek medical care immediately.
Patient knowledge on signs of labor, measured by patient survey | assessed between 36 - 42 weeks' gestation
  A count variable that measures the number of signs of labor a woman lists without being prompted.
Patient knowledge on breastfeeding, measured by patient survey | assessed between 36 - 42 weeks' gestation
  A binary variable that measures whether a woman correctly identifies the best time to start breastfeeding after delivery
Use of prenatal supplements, measured by patient survey | assessed between 36 - 42 weeks' gestation
  a binary variable that measures whether a woman is taking iron and folic acid supplementation tablets or prenatal supplement that contains iron and folic during her pregnancy
Birth preparation, measured by patient survey | assessed between 36 - 42 weeks' gestation
  a count variable that measures the total number of things a woman has done to prepare for her delivery
Institutional delivery, measured by patient survey | assessed between 7 - 8 weeks postpartum
  a binary variable that measures whether a woman delivered her baby in a hospital or health clinic/center
Exclusive breastfeeding, measured by patient survey | assessed between 7 - 8 weeks postpartum
  a binary variable that measures whether a baby is exclusively fed with breast milk
Sleep safety, measured by patient survey | assessed between 7- to 8-week postpartum
  A binary variable that measures weather a woman puts her baby to sleep in the safest position at night
Interaction with newborn, measured by patient survey | assessed between 7- to 8-week postpartum
  A binary variable that measures weather a woman spoke or sang to the baby in the past 24 hours
Patient self-efficacy in care-seeking during last antenatal care visit, measured by patient survey | assessed between 36 - 42 weeks' gestation
  a binary variable that measures whether a woman feels that she could ask healthcare workers at her last antenatal care visit any question she had about her pregnancy.
Patient self-efficacy in care-seeking during pregnancy and delivery, measured by patient survey | assessed between 7- to 8-week postpartum
  an ordinal variable that measures to what extent a woman feels she can get her questions about her health answered during pregnancy and delivery.
Timeliness of care, measured by delivery observation | assessed from patient arrival to up to 1 hour post the delivery of the placenta approximately 6 months after intervention initiation
  A continuous variable indicating delays in essential actions providers should perform, including time between facility arrival and first contact with health care worker, time between delivery and provision of uterotonic, time between delivery and breastfeeding initiation, and time between delivery and first maternal exam after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Cohen, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Margaret A McConnell, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Innovations for Poverty Actions, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
After manuscript publication, fully de-identified data may be shared with researchers upon request.

REFERENCES:
- [Background] Tripathi V, Stanton C, Strobino D, Bartlett L. Development and Validation of an Index to Measure the Quality of Facility-Based Labor and Delivery Care Processes in Sub-Saharan Africa. PLoS One. 2015 Jun 24;10(6):e0129491. doi: 10.1371/journal.pone.0129491. eCollection 2015. PMID 26107655
- [Background] Mbindyo PM, Blaauw D, Gilson L, English M. Developing a tool to measure health worker motivation in district hospitals in Kenya. Hum Resour Health. 2009 May 20;7:40. doi: 10.1186/1478-4491-7-40. PMID 19457237
- [Background] Berger BO, Strobino DM, Mehrtash H, Bohren MA, Adu-Bonsaffoh K, Leslie HH, Irinyenikan TA, Maung TM, Balde MD, Tuncalp O. Development of measures for assessing mistreatment of women during facility-based childbirth based on labour observations. BMJ Glob Health. 2021 Aug;5(Suppl 2):e004080. doi: 10.1136/bmjgh-2020-004080. PMID 34362791
- [Derived] Vatsa R, Chang W, Akinyi S, Little S, Gakii C, Mungai J, Kahumbura C, Wickramanayake A, Rajasekharan S, Cohen J, McConnell M. Impact evaluation of a digital health platform empowering Kenyan women across the pregnancy-postpartum care continuum: A cluster randomized controlled trial. PLoS Med. 2025 Feb 3;22(2):e1004527. doi: 10.1371/journal.pmed.1004527. eCollection 2025 Feb. PMID 39899612